CLINICAL TRIAL: NCT05932498
Title: Peri-capsular Nerve Group Block and Quadratus Lumborum Block for Hip Arthroplasty: A Randomized Controlled Trial
Brief Title: Peri-capsular Nerve Group (PENG) Block and Quadratus Lumborum Block for Hip Arthroplasty
Acronym: PENG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Po-Kai Wang, Director, Division of Pain Management, Department of Anesthesiology, Hualien Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB108-235-A
Record Dates: First submitted 2023-05-07; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Post Operative Pain
Keywords: postoperative pain; nerve block; regional analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: one group is that participants receive PENG block and another group is that participants receive QL block for postoperative pain control.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will not know which group they are in. Care provider, investigator, and outcomes assessor does not know which block participants will receive. The anesthesiologists who perform the blocks are not care provider, investigator, or outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG group (Experimental): Participants with PENG block
  Interventions: Procedure: Hip surgery
- QL group (Active Comparator): Participants with QL block
  Interventions: Procedure: Hip surgery

INTERVENTIONS:
Procedure: Hip surgery — Ultrasound-guided PENG block was administered to patients undergoing hip surgery intraoperatively.
  OR
  Ultrasound-guided QL block was administered to patients undergoing hip surgery intraoperatively.

SUMMARY:
The goal of this randomized controlled clinical trial is to compare peri-capsular nerve group (PENG) block and quadratus lumborum (QL) block in participants who receive hip arthroplasty. The main question aims to answer is comparing the pain score among participants who receive PENG or QL block.

Participants will be randomized and assigned into two groups. Participants will receive a PENG block in the PENG group and receive a QL block in the QL group. After participants receive hip arthroplasty, the investigators will compare the two groups to see if there is a difference of pain score, postoperative opioid consumption, sensation and motor function after nerve blocks, progress of functional recovery in lower limbs, intraoperative and postoperative complications.

DETAILED DESCRIPTION:
Hip joint surgery is a common orthopedic procedure that effectively improves patients' quality of life and functional status. However, postoperative pain is a common issue that can affect patients' activity, increase the risk of venous thromboembolism due to venous stasis, and prolong recovery time, hospital stay, and expenses. Therefore, controlling postoperative pain after hip joint surgery is crucial to reduce its side effects. Nerve block is one of the methods for postoperative pain management after hip joint surgery and has been proven effective in reducing pain levels, decreasing opioid use, and its side effects.

Traditionally, the quadratus lumborum nerve block (QL block) is used for pain relief during abdominal surgery, but it can also be used for lower limb surgery due to its extensive application. Compared to other nerve blocks, QL block may provide better postoperative pain relief, have less impact on hip joint activity and quadriceps muscle contraction, and reduce opioid use and hospital stay.

The peri-capsular nerve group block (PENG block) is another nerve block technique performed by injecting anesthetic analgesics around the hip joint capsule using ultrasound and blocking surrounding nerves with a larger dose. In a clinical study, PENG block significantly reduced static and dynamic pain scores in five patients with femoral neck fractures after 30 minutes of the nerve block. PENG block has advantages in injection and identification of anatomical structures compared to QL block, but their analgesic effects have not been directly compared. Therefore, clinical trials of both techniques are needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 20 years of age or older (including 20 years of age).
* Non-emergency hip arthroplasty surgery.
* Able to understand and cooperate with preoperative and postoperative data collection.
* Grade one to three in the American Society of Anesthesiologists (ASA) physical status classification.

Exclusion Criteria:

* Under 20 years of age.
* A known allergy to the study medication (ropivacaine).
* Liver cirrhosis classified as Child Pugh Score C.
* Dementia or mental illness.
* Unable to assess their own pain level.
* Patients who have been using opioid drugs for a prolonged period.
* Having a history of drug or alcohol abuse within the last 6 months.
* Having serious illness and at a risk of imminent mortality.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Comparing pain scores between the PENG and QL groups immediately after surgery | 10 minutes after surgery
  Pain scores were assessed using a standard Visual Analog Scale (VAS), where a rating of 0 indicated the absence of pain, while a score of 10 denoted the presence of the most severe pain.
Comparing pain scores between the PENG and QL groups at the 1-hour postoperative mark | at the 1-hour postoperative mark
  Pain scores were assessed using a standard Visual Analog Scale (VAS), where a rating of 0 indicated the absence of pain, while a score of 10 denoted the presence of the most severe pain.
Comparing pain scores between the PENG and QL groups at the 12-hour postoperative mark | at the 12-hour postoperative mark
  Pain scores were assessed using a standard Visual Analog Scale (VAS), where a rating of 0 indicated the absence of pain, while a score of 10 denoted the presence of the most severe pain.
Comparing pain scores between the PENG and QL groups at the 24-hour postoperative mark | at the 24-hour postoperative mark
  Pain scores were assessed using a standard Visual Analog Scale (VAS), where a rating of 0 indicated the absence of pain, while a score of 10 denoted the presence of the most severe pain.
Comparing pain scores between the PENG and QL groups at the 48-hour postoperative mark | at the 48-hour postoperative mark
  Pain scores were assessed using a standard Visual Analog Scale (VAS), where a rating of 0 indicated the absence of pain, while a score of 10 denoted the presence of the most severe pain.

SECONDARY OUTCOMES:
Postoperative opioid consumption | at the 12-, 24-, 48-hours after surgery
  Comparing the amount of parenteral opioids administered for rescue purposes as Morphine Milligram Equivalents (MME) between the PENG and QL groups at various postoperative time intervals.
The quadriceps strength on surgical side | at the 0-, 1-, 12-, 24-, 48-, and 72-hours after surgery
  After performing PENG or QL blocks, the investigators assessed and compared the strength of the quadriceps muscles on the side that underwent hip surgery using Manual Muscle Testing (MMT) scores. MMT involves assigning scores to assess the patients' quadriceps muscle strength, ranging from 0 (no activation) to 5 (activation against resistance).
Time to independently sit at the edge of the bed after surgery | From the date of hip surgery until the patient achieves independent sitting at the edge of the bed, with a maximum follow-up period of 7 days
  Sitting at the edge of the bed is a functional milestone that reflects the patient's progress toward regaining mobility and independence in activities of daily living.
  The duration required to achieve sitting at the edge of the bed was measured in terms of the number of days following the surgery.
Time to stand up after surgery | From the date of hip surgery until the patient achieves standing up, with a maximum follow-up period of 7 days
  Standing up indicates the patient's ability to bear weight on the affected hip joint and engage in activities such as walking, transferring, and performing daily tasks after hip surgery.
  The duration required to achieve standing up was measured in terms of the number of days following the surgery.
Time to walk with the aid of walking devices after surgery | From the date of hip surgery until the patient achieves walking with the aid of walking devices, with a maximum follow-up period of 7 days
  Walking with the aid of walking devices reflects the patient's ability to regain mobility and independence in walking, even if patients require assistance or support from these devices.
  The duration required to achieve walking with the aid of walking devices was measured in terms of the number of days following the surgery.
Perioperative blood loss and blood transfusion | During the surgery and over the three-day postoperative period
  The investigators documented the amount of blood loss and the need for blood transfusion both during the surgery and in the postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Po-Kai Wang, MD, PhD, Principal Investigator — Hualien Tzu Chi General Hospital
Locations (1):
- Po-Kai Wang, Hualien City, Hualien, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Min BW, Kim Y, Cho HM, Park KS, Yoon PW, Nho JH, Kim SM, Lee KJ, Moon KH. Perioperative Pain Management in Total Hip Arthroplasty: Korean Hip Society Guidelines. Hip Pelvis. 2016 Mar;28(1):15-23. doi: 10.5371/hp.2016.28.1.15. Epub 2016 Mar 31. PMID 27536639
- [Background] Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID 28154824
- [Background] La Colla L, Ben-David B, Merman R. Quadratus Lumborum Block as an Alternative to Lumbar Plexus Block for Hip Surgery: A Report of 2 Cases. A A Case Rep. 2017 Jan 1;8(1):4-6. doi: 10.1213/XAA.0000000000000406. PMID 28036319
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657